CLINICAL TRIAL: NCT01276691
Title: Effect of Aspirin on Hemostatic and Vascular Function After Live Fire Fighting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gavin Horn, Senior Research Scientist, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: AsprinFire2011
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Risk Factor; C.Medical Procedure; Vascular, Functional or Late; Electrolyte and Fluid Balance Conditions
Keywords: Vascular function; Inflammation; Oxidative stress; Hemostatic balance; Aspirin; Firefighting
MeSH Terms: conditions — Inflammation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acute, Aspirin (Active Comparator): 81 mg asprin provided 30 minutes prior to firefighting- Acute single dosage
  Interventions: Drug: 81 mg enteric coated aspirin
- Acute, Placebo (Placebo Comparator): Acute single dosage of placebo provided 30 minutes prior to firefighting
  Interventions: Drug: 81 mg enteric coated aspirin
- Chronic, Aspirin (Active Comparator): 81 mg asprin provided prior to firefighting- 14 day dosage
  Interventions: Drug: 81 mg enteric coated aspirin
- Chronic, Placebo (Placebo Comparator): 14 day dosage of placebo provided prior to firefighting
  Interventions: Drug: 81 mg enteric coated aspirin

INTERVENTIONS:
Drug: 81 mg enteric coated aspirin — 81 mg enteric coated aspirin will be provided both as an acute dosage immediately prior to firefighting (1 hour pre-activity) and as a 14 day dosage prior to firefighting
  Other Names: aspirin

SUMMARY:
The investigators hypothesize that

1. an acute treatment of low-dose aspirin will lead to a) decreased resting platelet activation, platelet aggregation, and clotting potential, b) increased fibrinolytic potential following fire fighting, c) no significant effect on endothelial function or arterial stiffness versus the placebo condition.
2. chronic treatment with low-dose aspirin will lead to a) decreased resting and fire fighting induced platelet activation, platelet aggregation, clotting potential, b) increased fibrinolytic potential, and c) increased endothelial function and decreased arterial stiffness in response to live fire fighting versus the placebo condition.
3. short-term fire fighting activity will result in: a) a reduction in arterial function (reduced endothelial function, increased augmentation index and an attenuated arterial stiffness response); b) a disruption in hemostasis that is characterized by an increase in platelet number and function, an increased coagulatory potential and altered fibrinolytic potential; and c) an elevation in procoagulatory cytokines, systemic inflammation, monokine chemoattractant protein, and matrix metalloproteinases.

ELIGIBILITY:
Inclusion Criteria:

* Male firefighters (career and volunteer), medically cleared by home fire department.
* Ages 40 - 60
* Completion of a yearly period medical evaluation based on NFPA 1582 within the past 12 months or an evaluation by an occupational medical group through this study.

Exclusion Criteria:

* Over 60 or under 40 years of age.
* Not a firefighter.
* Individuals at risk for developing gastrointestinal (GI) complications while on aspirin therapy due to a combination of the following: smoking; concurrent NSAID, steroid, Clopidogrel, or Warfarin therapy; history of upper GI complications; history of renal impairment; history of elevated serum creatinine; hypertension; and cardiac failure.
* Individuals with cases of allergy or asthma, intolerance, and recurrent vascular events.
* Individuals taking statins.
* Individuals who are currently taking aspiring regularly.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Vascular function | Less than 60 minutes before initiating firefighting activity
  Vascular function will be assessed via pulse wave analysis, pulse wave velocity, carotid artery compliance, beta stiffness index, forearm rsistance artery vasodilatory capacity, and brachial artery blood flow.
Hemostatic balance | Less than 60 minutes before initiating firefighting activity
  Blood samples will be collected by a trained phlebotomist from the antecubital vein directly into vacutainers with little or no stasis using a 21-gauge needle. Samples will be used to quantify platetlet number and function, fibrinogen, prothrombin and partial thromboplastin time, t-PA and PAI-1 activities and antigen
Inflammatory and Oxidative Stress markers | Less than 60 minutes before initiating firefighting activity
  CRP,Intercellular adhesion molecule (ICAM)-1, IL-6, MMP-9, TIMP-1, TIMP-2,8-iso-prostaglandin F2a, soluble P-selectin
Vascular function | Less than 60 minutes after completing 20 minutes of firefighting activity
  Vascular function will be assessed via pulse wave analysis, pulse wave velocity, carotid artery compliance, beta stiffness index, forearm rsistance artery vasodilatory capacity, and brachial artery blood flow.
Hemostatic balance | Less than 60 minutes after completing 20 minutes of firefighting activity
  Blood samples will be collected by a trained phlebotomist from the antecubital vein directly into vacutainers with little or no stasis using a 21-gauge needle. Samples will be used to quantify platetlet number and function, fibrinogen, prothrombin and partial thromboplastin time, t-PA and PAI-1 activities and antigen
Inflammatory and Oxidative Stress markers | Less than 60 minutes after completing 20 minutes of firefighting activity
  CRP,Intercellular adhesion molecule (ICAM)-1, IL-6, MMP-9, TIMP-1, TIMP-2,8-iso-prostaglandin F2a, soluble P-selectin

CONTACTS AND LOCATIONS:
Overall Officials: Gavin P Horn, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- Illinois Fire Service Institute, Champaign, Illinois, United States

REFERENCES:
- [Derived] Smith DL, Friedman NMG, Bloom SI, Armero WL, Pence BD, Cook MD, Fernhall B, Horn GP, Woods J. Firefighting Induces Acute Inflammatory Responses that are not Relieved by Aspirin in Older Firefighters. J Occup Environ Med. 2019 Jul;61(7):617-622. doi: 10.1097/JOM.0000000000001626. PMID 31090673
- [Derived] Lane-Cordova AD, Ranadive SM, Yan H, Kappus RM, Sun P, Bunsawat K, Smith DL, Horn GP, Ploutz-Snyder R, Fernhall BO. Effect of Aspirin Supplementation on Hemodynamics in Older Firefighters. Med Sci Sports Exerc. 2015 Dec;47(12):2653-9. doi: 10.1249/MSS.0000000000000713. PMID 26057939
- See also: Illinois Fire Service Institute home page — http://www.fsi.illinois.edu